CLINICAL TRIAL: NCT06693999
Title: Automated Coping Interventions to Enhance Physical Activity Among Stroke Survivors
Brief Title: Just In Time Intervention to Enhance Physical Activity Among Stroke Survivors
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Ramin Zand, Professor of Neurology, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00025868
Record Dates: First submitted 2024-11-15; First posted 2024-11-19 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Stroke
Keywords: Stroke; Physical Activity; Wearable tracker; Smart Phone
MeSH Terms: conditions — Stroke; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adult stroke Survivors (Other): This arm consists of stroke survivors with specified inclusion/exclusion criteria who will receive goal reminders and motivational, in addition to coping messages through Google Pixel Watches.
  Interventions: Device: Google-Pixel Watch 3; Behavioral: Exercise prompts

INTERVENTIONS:
Device: Google-Pixel Watch 3 — The participant will wear Google-Pixel Watch 3 for at least 10 hours during the 3-month intervention and will receive goal reminders and motivational and coping messages through those watches. At baseline and after 3-months intervention, demographics (standard questionnaire pertaining to subjects' age, sex, race, education and income), technology literacy (eHealth Literacy Scale pertaining to subjects' ability to perform a number of tasks such as turning on the device, using internet and communication), and wearables affinity (pertains to how the subject currently uses wearable in their daily living tasks) will be measured.
Behavioral: Exercise prompts — The participants will receive goal reminders.

SUMMARY:
A 3-month single-arm pilot trial to evaluate the feasibility of an automated and individualized coping intervention among stroke survivors.

ELIGIBILITY:
Inclusion Criteria:

1. Adult Patients Diagnosed with Stroke: Participants must be adults (age ≥ 18) who have been clinically diagnosed with a stroke between 3 months and 3 years.
2. Community-Dwelling: Participants should be living independently in the community rather than in institutional settings such as nursing homes or hospitals.
3. Independently Mobile: Participants must be able to walk without any aid or assistance, corresponding to a modified Rankin Scale (mRS) score of 0-2.
4. Physically Inactive: Participants should have engaged in less than 10 minutes of moderate-to-vigorous physical activity (MVPA) in the past week.
5. Internet Access: Participants must have access to the Internet for at least a few hours every day.
6. Medically Cleared to participate: Before enrollment, participants must obtain medical clearance to ensure they are fit to participate in the study.

Exclusion Criteria:

1. Participating in Another Research Project Involving Physical Activity: To avoid potential confounding variables that could affect the study's outcomes.
2. Planning to Move or Have Surgery in the Next 6 Months: Participants who plan to move or undergo surgery within the next six months may face disruptions that could affect their ability to complete the study.
3. Cognitive Impairment: Cognitive impairment can affect a participant's ability to understand and follow study protocols, which is crucial for informed consent and reliable data collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants retained | 3 months
  The number of participants who remain in the study until its conclusion.

SECONDARY OUTCOMES:
Number of subjects recruited for the study | 3 months
  This measures how effectively participants are being enrolled in the study.
Number of hours devices were worn | 3 months
  Number of hours device were worn by the subjects.
Number of prompts | 3 months
  This refers to the number of prompts responded by participants throughout the study duration.

OTHER OUTCOMES:
Weekly Goal Adherence | 3 months
  Number of weekly physical activity goals met by the participants throughout the study.
Minutes of Physical Activity | 3 months
  The total time spent in light, moderate and vigorous physical activity during the study period. Light, moderate and vigorous physical activity are defined based on subjects' maximal heart rate. Maximal Heart Rate (MHR) = 220 - subject's age. Light is defined as 30-50% of MHR, moderate intensity as 50-75% of MHR and vigorous intensity as 70-85% of MHR according to American Heart Association. For instance, a 50-year-old subject's maximum heart rate would be 220 - 50 = 170. For the subject to be doing moderate intensity, their heart rate should be in between 85-127 and 119-144 to perform vigorous physical activity.

IPD SHARING:
Plan to Share IPD: Undecided